CLINICAL TRIAL: NCT01651806
Title: Weighted Versus Uniform Dose of Tranexamic Acid in Patients Undergoing Primary, Knee Arthroplasty, a Randomized-clinical Trial.
Brief Title: Weighted Versus Uniform Dose of Tranexamic Acid in Patients Undergoing Primary, Knee Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brett Levine, MD, Assistant Professor and Associate Residency Director, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12021202
Record Dates: First submitted 2012-05-01; First posted 2012-07-27 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis; Intraoperative Bleeding
Keywords: Blood loss; transfusion rates; complications
MeSH Terms: conditions — Osteoarthritis; Blood Loss, Surgical; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Females receiving a uniform dose of TA (Active Comparator): Women receiving a single dose of 1 gram of TA--includes all women that will get 1 gram dose of the TA during surgery. Postop outcomes wil be measured for comparison, including hemoglobin, hematocrits and blood loss.
  Interventions: Drug: Females receiving a uniform dose of TA
- Weighted dose of TA in female patients (Active Comparator): Female patients receiving a weighted dose of TA. Will include all women that will get a weighted dose of the TA during surgery. Postop outcomes wil be measured for comparison, including hemoglobin, hematocrits and blood loss.
  Interventions: Drug: Females Tranexamic Acid weighted dose
- Tranexamic acid weighted dose male (Active Comparator): Male patients randomized to the weighted dose of TA. Postop outcomes wil be measured for comparison, including hemoglobin, hematocrits and blood loss.
  Interventions: Drug: Males Weighted Dose TA
- Uniform single dose TA male patient (Active Comparator): Male patients receiving a single dose (1gram) of TA during TKA. Includes all men that will get 1 gram dose of the TA during surgery. Postop outcomes wil be measured for comparison Postop outcomes wil be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Interventions: Drug: Tranexamic Acid standard dose
- Historical Cohort (No Intervention): 25 patients with no TA use in their surgical history.
  A control group was established from a historical cohort of primary TKAs performed by the senior author (BL), none of which received TA. The most relevant Pubmed ID would be 24997651.

INTERVENTIONS:
Drug: Tranexamic Acid standard dose — Uniform 1 gram dosing
  Other Names: Male TA
  Arms: Uniform single dose TA male patient
Drug: Females Tranexamic Acid weighted dose — Weighted dose--20mg/kg of the drug will be given
  Other Names: TA
  Arms: Weighted dose of TA in female patients
Drug: Females receiving a uniform dose of TA — Patients will receive a uniform 1 gm dose of tranexamic acid prior to tourniquet release during a primary TKA.
  Other Names: Tranexamic Acid
  Arms: Females receiving a uniform dose of TA
Drug: Males Weighted Dose TA — Weighted dose--20mg/kg of the drug will be given
  Other Names: Transexamic Acid
  Arms: Tranexamic acid weighted dose male

SUMMARY:
Hypotheses: Primary - A weighted dose of 20 mg/kg of tranexamic acid will be more efficacious than a single uniform dose of 1 gram in primary total knee arthroplasty (TKA) cases. This includes having a greater impact on decreasing blood loss without increasing the occurrence of adverse thromboembolic events in patients undergoing primary, elective total knee arthroplasty.

Secondary - TA will decrease blood loss more effectively in women than in men undergoing this procedure.

DETAILED DESCRIPTION:
Overall Study Design

Study design and control methods:

This study is designed as a prospective, randomized, double-blinded controlled clinical trial to compare the effect of a single uniform 1 g dose of TA and a single weighted 20 mg/kg dose of tranexamic acid (TA).

Treatment group:

The subjects will be randomly assigned to the uniform dose group or weighted dose group at the time of the surgery via the opening of a randomly selected closed envelope. The patient and the independent reviewer will be blinded as to the dose of TA utilized during the surgery. This information will be linked to a confidential database for later review by the principal investigator.

Treatment allocation:

All eligible patients (i.e., meeting inclusion criteria and no exclusion criteria) will be treated and observed per the research protocol. All patients will maintain the right to refuse participation and receive a specific treatment of the study if desired.

Trial Population

Target population:

The target sample size is 60 patients of each of the uniform and weighted dose groups (120 total). There will be one actively enrolling surgeon (Dr. Brett Levine). The goal is to enroll a total of 120 subjects experiencing joint pain that warrants a TKA. The specific diagnosis for the joint pain will not direct the subjects' assignment or eligibility at the time of surgery. All 120 patients will be enrolled from the office of the primary investigator (Dr. Brett Levine). All indications for TKA will be included unless one of the exclusion criteria is met.

Results from randomized patients will be compared to a historical control arm that did not receive TA in their treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be male or female of any race
2. Ages 18-80 years old
3. Patients must be undergoing an elective, primary knee arthroplasty
4. Patients must be able to understand and willing to cooperate with study procedures
5. Patients must be able to provide written and verbal informed consent

Exclusion Criteria:

1. Allergy or intolerance to the study materials
2. History of a venous thromboembolic event being treated with life-long anticoagulation
3. Patients with a known congenital thrombophilia
4. Patients who have had a venous thromboembolic event within the 12 months preceding surgery
5. History of any substance abuse or dependence within the last 6 months
6. Failure in collecting a required data point during study
7. Those patients not indicated for knee replacement surgery including, pregnant women, those not cleared medically for the procedure and patients without significant radiographic evidence of degenerative joint disease.
8. Patient using autologous blood transfusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Belkin, BS, Study Director — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] Husted H, Blond L, Sonne-Holm S, Holm G, Jacobsen TW, Gebuhr P. Tranexamic acid reduces blood loss and blood transfusions in primary total hip arthroplasty: a prospective randomized double-blind study in 40 patients. Acta Orthop Scand. 2003 Dec;74(6):665-9. doi: 10.1080/00016470310018171. PMID 14763696
- [Background] Ralley FE, Berta D, Binns V, Howard J, Naudie DD. One intraoperative dose of tranexamic Acid for patients having primary hip or knee arthroplasty. Clin Orthop Relat Res. 2010 Jul;468(7):1905-11. doi: 10.1007/s11999-009-1217-8. Epub 2010 Jan 9. PMID 20063079

RESULTS

PARTICIPANT FLOW:
Groups:
- Female Uniform Single Dose TA Patient: Female patients receiving a single dose (1gram) of TA during TKA. Includes all female patients that will get 1 gram dose of the TA during surgery. Postop outcomes will be measured for comparison Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Uniform 1 gram dosing
- Female Weighted Dose TA Patient: Female patients receiving a weighted dose (20mg/kg) of TA during TKA. Postop outcomes will be measured for comparison Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Weighted 20mg/kg gram dosing
- Control: Historical cohort of primary TKAs performed by BL, none of which received TA.
  A control group was established from a historical cohort of primary TKAs performed by the senior author (BL), none of which received TA. The most relevant Pubmed ID would be 24997651.
- Male Uniform Single Dose TA Patient: Male patients receiving a single dose (1gram) of TA during TKA. Includes all male patients that will get 1 gram dose of the TA during surgery. Postop outcomes will be measured for comparison Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Uniform 1 gram dosing
- Male Weighted Dose TA Patient: Male patients receiving a weighted dose (20mg/kg) of TA during TKA. Postop outcomes will be measured for comparison Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Weighted 20mg/kg gram dosing
Period: Overall Study
Arm/Group | Female Uniform Single Dose TA Patient | Female Weighted Dose TA Patient | Control | Male Uniform Single Dose TA Patient | Male Weighted Dose TA Patient
Started | 13 | 12 | 25 | 7 | 8
Completed | 13 | 12 | 25 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Female Patients Receiving a Uniform Dose of TA: Female Patients receiving a single dose of 1 gram of TA--includes all patients that will get 1 gram dose of the TA during surgery. Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss.
  Patients will receive a uniform 1 gm dose of tranexamic acid prior to tourniquet release during a primary TKA.
- Female Weighted Dose of TA Patients: Female Patients receiving a weighted dose of TA. Will include all patients that will get a weighted dose of the TA during surgery. Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss.
  Tranexamic Acid weighted dose: Weighted dose--20mg/kg of the drug will be given
- Control: Historical cohort of primary TKAs performed by senior author, none of which received TA.
- Male Patients Receiving a Uniform Dose of TA: Male Patients receiving a single dose of 1 gram of TA--includes all patients that will get 1 gram dose of the TA during surgery. Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss.
  Patients will receive a uniform 1 gm dose of tranexamic acid prior to tourniquet release during a primary TKA.
- Male Weighted Dose of TA Patients: Male Patients receiving a weighted dose of TA. Will include all patients that will get a weighted dose of the TA during surgery. Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss.
  Tranexamic Acid weighted dose: Weighted dose--20mg/kg of the drug will be given
- Total: Total of all reporting groups
Arm/Group | Female Patients Receiving a Uniform Dose of TA | Female Weighted Dose of TA Patients | Control | Male Patients Receiving a Uniform Dose of TA | Male Weighted Dose of TA Patients | Total
Number analyzed (Participants) | 13 | 12 | 25 | 7 | 8 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 15 | 4 | 3 | 35
  >=65 years | 5 | 7 | 10 | 3 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.26 (7.31) | 66.50 (9.65) | 62.40 (10.1) | 62.26 (7.31) | 66.50 (9.65) | 64.38 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 15 | 0 | 0 | 40
  Male | 0 | 0 | 10 | 7 | 8 | 25
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.10 (8.04) | 35.40 (8.50) | 36 (11.09) | 32.10 (8.04) | 35.40 (8.50) | 33.75 (8.436)
ASA [Mean (Standard Deviation); unit: Scores on a Scale] — American Society of Anesthesiologists (ASA) Score is a global score that assesses the physical status of patients before surgery.
  It is sometimed refereed to as ASA-PS, because it is a measure of 'physical status'.
  ASA 1 A normal healthy patient. ASA 2 A patient with mild systemic disease. ASA 3 A patient with severe systemic disease. ASA 4 A patient with severe systemic disease that is a constant threat to life. ASA 5 A moribund patient who is not expected to survive
  The ASA Score is a useful global measure of health.
  Scores on a Scale | 2.53 (0.6) | 2.26 (0.7) | 2.57 (0.5) | 2.53 (0.6) | 2.26 (0.7) | 2.395 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Primary Intra-operative Blood Loss
Description: Record intra-operative blood loss through drain output
Time Frame: Intra-operative, an average of 3 hours
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Female Uniform Single Dose TA Patient: Female patients receiving a single dose (1gram) of TA during TKA. Includes all patients that will get 1 gram dose of the TA during surgery. Postop outcomes will be measured for comparison Postop outcomes wil be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Uniform 1 gram dosing
- Control: Historical cohort of primary TKAs performed by BL, none of which received TA.
- Male Uniform Single Dose TA: Male patients receiving a single dose (1gram) of TA during TKA. Includes all patients that will get 1 gram dose of the TA during surgery. Postop outcomes will be measured for comparison Postop outcomes wil be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Uniform 1 gram dosing
- Male Weighted Dose TA Patient: Female patients receiving a weighted dose (20mg/kg) of TA during TKA. Postop outcomes will be measured for comparison Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Weighted 20mg/kg gram dosing
Arm/Group | Female Uniform Single Dose TA Patient | Female Weighted Dose TA Patient | Control | Male Uniform Single Dose TA | Male Weighted Dose TA Patient
Number analyzed (Participants) | 13 | 12 | 25 | 7 | 8
mL | 100.00 (31.69) | 65.00 (8.50) | 142.80 (197) | 100.00 (31.69) | 65.00 (8.50)

2. Primary Outcome: Document Incidences of DVT and Other Thromboembolic Events.
Description: DVT = Deep Venous thrombosis
  Patients were assessed every 12 hours for development of pain within the lower extremity. Any reported muscle pain was evaluate with a bedside venous ultrasound by an ultrasound technician.
Time Frame: 1 year
Measure: Number; unit: Events
Groups:
- Male Weighted Dose TA: Male patients receiving a weighted dose (20mg/kg) of TA during TKA. Postop outcomes will be measured for comparison Postop outcomes will be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Weighted 20mg/kg gram dosing
Arm/Group | Female Uniform Single Dose TA Patient | Female Weighted Dose TA Patient | Control | Male Uniform Single Dose TA | Male Weighted Dose TA
Number analyzed (Participants) | 13 | 12 | 25 | 7 | 8
Events | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Male Uniform Single Dose TA Patient: Male patients receiving a single dose (1gram) of TA during TKA. Includes all patients that will get 1 gram dose of the TA during surgery. Postop outcomes will be measured for comparison Postop outcomes wil be measured for comparison, including hemoglobin, hematocrits and blood loss. Patients will be randomized into one of these two groups.
  Tranexamic Acid standard dose: Uniform 1 gram dosing
Arm/Group | Female Uniform Single Dose TA Patient | Female Weighted Dose TA Patient | Control | Male Uniform Single Dose TA Patient | Male Weighted Dose TA
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/12 | 0/25 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 1/12 | 10/25 | 0/7 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Female Uniform Single Dose TA Patient (N=13) | Female Weighted Dose TA Patient (N=12) | Control (N=25) | Male Uniform Single Dose TA Patient (N=7) | Male Weighted Dose TA (N=8)
Symptomatic DVT (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Female Uniform Single Dose TA Patient (N=13) | Female Weighted Dose TA Patient (N=12) | Control (N=25) | Male Uniform Single Dose TA Patient (N=7) | Male Weighted Dose TA (N=8)
Blood Transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 10 (10) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No